CLINICAL TRIAL: NCT02233231
Title: Smoking Young Asthmatics: Change of Inflammation During Tobacco Cessation and Steroid Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vibeke Backer (Other)
Responsible Party: Sponsor-Investigator, Vibeke Backer, MD, DMSCI, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Young smoking asthmatics
Record Dates: First submitted 2013-03-18; First posted 2014-09-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2014-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): Varenicline 0,5 mg x 1 day 1-3 Varenicline 0,5 mg x 2 day 4-6 Varenicline 2 mg x 1 day 7 to week 12
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Placebo tablets equivalent to IMP.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline 2 mg x 1 day 7 to week 12
  Other Names: Placebo
  Arms: Varenicline
Drug: Placebo — similar tabl
  Other Names: Varenicline
  Arms: Placebo

SUMMARY:
This is a study describing changes in inflammation of the airways in asthmatics before and after smoking cessation and steroid treatment.

DETAILED DESCRIPTION:
84 smoking asthmatics will be included. 50% will be treated with varenicline and 50% with placebo tablets for 12 weeks. All will be treated with inhaled steroid for 12 weeks.

Study period: About 26 weeks including asthma screening. 4 visits will be performed. Inflammation will be described through sputum induction, and several other pulmonary medical tests will be performed, including NO, methacholine, spirometry, CO, blood samples, skin prick test and asthma questionaires.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic symptoms during the last year and at least one criterion of the below:

1. current FEV1-increase of minimum 12% after b2-agonist,
2. positiv Methacholintest,
3. Day-to-day FEV1-variation of at least 20% during a two-week period.
4. Positive mannitol test.

Furthermore, all of the below inclusion criteria:

* At least 10 packyears
* At least 10 cigarettes per day within the last year
* Age 18-40 years

Exclusion Criteria:

1. Asthmatics who have been treated with inhaled corticosteroids (ICS), systemic corticosteroids, leukotrien-antagonists (LTA), long-lasting b2-agonists, anticholinergic medicine or varenicline within the last 3 months
2. Lower respiratory tract infections, including pneumonia, within the last 6 weeks.
3. Patients suffering from other chronic respiratory disease than asthma, such as sarcoidosis and COPD will also be excluded.
4. Pregnant and nursing women will be excluded as well as women planning pregnancy during the study period.
5. A history of allergy towards study drugs will lead to exclusion.

Patients who during the study period develop lower respiratory infections or due to severe uncontrolled asthma receive treatment with any of the above listed types of medicine will be excluded. Patients who are diagnosed with other chronic respiratory disease than asthma during the study period will also be excluded, as well as patients who during the study period require more asthma medicine than the planned study medication.

Any participant who wishes to leave the study, for any reason, including unacceptable side-effects, during the study period will be excluded, as well as anyone who wants to withdraw their recorded data from the project after the study period has ended.

In case of unacceptable side-effects to varenicline resulting in immediate cessation of treatment with this drug, the participant will continue visits unchanged, but he/she will be excluded from the calculations of tobacco cessation succes-rate. However, varenicline cessation up to 4 weeks after treatment start with varenicline will result in exclusion and replacement of the participant.

Cessation of treatment with budesonide will result in exclusion from the rest the study. The person will not be replaced. The data recorded from the participant until the last visit before cessation will be used.

Allergic reactions towards study drugs will result in immediate cessation of the drug, and possible exclusion, as described in the above.

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in sputum eosinophile-% from >1% to normal or neutrophile-% from >61% to normal, from baseline (week 0) to week 12. | Time frame for primary outcome: 0-12 weeks (total study duration 24 weeks)
  Power calculations are based on changes during 0-12 weeks.
  The total study includes primary outcome measurements at:
  Visit 1: Week 0, Visit 2: Week 6, Visit 3: Week 12, Visit 4: Week 24

SECONDARY OUTCOMES:
Change in methacholine hyperresponsiveness by two dosis steps, from baseline (week 0) to week 12. | Time frame for secondary outcome: 0-12 weeks
  The secondary outcome are measured at:
  Visit 1: Week 0, Visit 2: Week 6, Visit 3: Week 12, Visit 4: Week 24

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273